CLINICAL TRIAL: NCT07180511
Title: A Multicenter, Randomized, Parallel, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of QY201 Tablets in Subjects With Moderate to Severe Atopic Dermatitis.
Brief Title: A Phase III Clinical Study of QY201 Tablet in Subjects With Moderate to Severe Atopic Dermatitis.
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: E-nitiate Biopharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QY201-301
Record Dates: First submitted 2025-09-10; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- QY201 placebo tablet (Placebo Comparator): Using QY201placebo tablet twice daily for 16 weeks
  Interventions: Drug: 10mg QY201 Placebo tablet; Drug: 20mg QY201 Placebo tablet
- 20mg QY201 tablet (Experimental): Using 20mg QY201 tablet twice daily for 52 weeks
  Interventions: Drug: 10mg QY201 Placebo tablet; Drug: 20mg QY201 tablet
- 10mg QY201 tablet (Experimental): Using 10mg QY201 tablet twice daily for 52 weeks
  Interventions: Drug: 20mg QY201 Placebo tablet; Drug: 10mg QY201 tablet

INTERVENTIONS:
Drug: 10mg QY201 Placebo tablet — 10mg QY201 Placebo tablet
  Arms: 20mg QY201 tablet; QY201 placebo tablet
Drug: 20mg QY201 Placebo tablet — 20mg QY201 Placebo tablet
  Arms: 10mg QY201 tablet; QY201 placebo tablet
Drug: 10mg QY201 tablet — 10mg QY201 tablet
  Arms: 10mg QY201 tablet
Drug: 20mg QY201 tablet — 20mg QY201 tablet
  Arms: 20mg QY201 tablet

SUMMARY:
To evaluate the efficacy of QY201 tablets in the treatment of adult patients with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to communicate well with the investigator, fully understand the trial's purpose, nature, methods, and potential adverse reactions, voluntarily agrees to participate as a subject, understands and complies with all requirements of the study, and signs the ICF before any study procedures begin;
2. At the time of signing the ICF, the subject is between 18 and 75 years of age (inclusive), regardless of gender;
3. Has a history of AD for at least 1 year at screening and meets the Hanifin-Rajka diagnostic criteria (see Appendix 1) at screening;
4. Meets the criteria for moderate-to-severe AD at both screening and baseline (all 4 criteria must be met):

   * vIGA-AD score ≥3 at screening and baseline (see Appendix 2);
   * EASI score ≥16 at screening and baseline (see Appendix 3);
   * BSA ≥10% at screening and baseline (see Appendix 4);
   * Weekly average of daily PP-NRS score ≥4 at baseline (see Appendix 6); [Note] The weekly average of the daily PP-NRS score at baseline will be calculated based on the scores recorded daily during the 7 consecutive days prior to baseline. If there are fewer than 7 days of daily PP-NRS scores during the 7 consecutive days prior to baseline, scores from at least 4 days must be used for the calculation. If there are fewer than 4 days, randomization should be postponed, but must not exceed the maximum screening period of 35 days.
5. Within 6 months prior to screening, there is a documented history indicating an inadequate response or intolerance to topical treatments such as TCS and/or TCI; or a documented history indicating the need for systemic therapy (e.g., systemic corticosteroids, conventional immunosuppressants, biologics, Janus kinase [JAK] inhibitors, etc.) to control the disease; [Note] Inadequate response is defined as failure to achieve disease remission or maintain a low disease activity state despite using mid-potency or potent TCS for at least 4 weeks or superpotent TCS for at least 2 weeks as prescribed, or using TCI for at least 4 weeks. Intolerance is defined as worsening of skin lesions after 1-2 weeks of topical treatment, or the occurrence of discomfort including pain, burning, or uncomfortable sensations following drug use.
6. The subject is able and willing to regularly use a mild, additive-free emollient at least twice daily for at least 7 consecutive days prior to randomization and to continue its use throughout the study period.
7. The subject (including their partner) agrees to have no pregnancy plans from the time of signing the ICF until 3 months after the last dose and voluntarily adopts effective contraceptive measures ;

   * Male subjects: Must agree not to donate sperm during the study and for 3 months after the last study drug administration.
   * Female subjects:

     * Women of childbearing potential: Must have a negative serum human chorionic gonadotropin (HCG) test during the screening period and must not be breastfeeding.
     * Women without childbearing potential: Permanently sterilized (e.g., bilateral oophorectomy, bilateral salpingectomy, hysterectomy) or postmenopausal (defined as cessation of menstruation for at least 12 months with other pathological causes excluded; for women under 60 years old, serum follicle-stimulating hormone [FSH] level >40 IU/L must be confirmed).

Exclusion Criteria:

Have used any of the following drugs/treatments within the specified time frames:

1. Previously participated in any clinical trial of QY201 tablets;
2. Used the following systemic treatments within 12 weeks before baseline (or 5 half-lives, whichever is longer):

   * Small molecule targeted drugs: JAK inhibitors (e.g., Ruxolitinib, Tofacitinib, Baricitinib, Upadacitinib, Abrocitinib), etc.;
   * Macromolecular biologics: such as Dupilumab, etc.;
3. Used the following systemic treatments within 4 weeks before baseline (or 5 half-lives, whichever is longer):

   * Systemic immunosuppressants/immunomodulatory drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate mofetil, interferon gamma, azathioprine, methotrexate, etc.);
   * Phototherapy (e.g., ultraviolet B [UVB], psoralen + ultraviolet A [PUVA], etc.), including indoor tanning;
   * Systemic traditional Chinese herbal medicines or proprietary Chinese medicines that may affect efficacy evaluation;
   * Other systemic drugs for treating AD;
4. Used topical JAK inhibitors for local treatment within 4 weeks before baseline; used the following local treatments within 1 week before baseline:

   * TCS;
   * TCI;
   * Topical phosphodiesterase-4 (PDE-4) inhibitors;
   * Topical traditional Chinese medicine preparations or local herbal baths that may affect efficacy evaluation;
   * Other local drugs for treating AD;
5. Received allergen-specific immunotherapy within 6 months before baseline;
6. Used strong inhibitors or inducers of cytochrome P450 3A enzyme (CYP3A) within 2 weeks before baseline (see Appendix 9);
7. Used long-acting anticoagulants (e.g., warfarin, clopidogrel, etc.) within 4 weeks before baseline or required continuous use of anticoagulant therapy (except aspirin ≤100 mg/day);
8. Planned to receive live vaccines or live attenuated vaccines within 4 weeks before baseline; or expected to require live vaccines or live attenuated vaccines during the study period (including at least 4 weeks after the last dose of the investigational product);
9. Participated in and used any investigational drug within 4 weeks (or 5 half-lives, whichever is longer) before baseline, or participated in and used any medical device in a clinical trial within 3 months;

   Have any of the following medical histories or abnormalities:
10. Other skin comorbidities that, in the investigator's assessment, may interfere with the study evaluation, aside from AD;
11. History of disseminated herpes zoster (a single episode) or disseminated herpes simplex (a single episode), or recurrent (≥2 episodes) localized herpes zoster;
12. Diagnosed or suspected active tuberculosis, latent untreated tuberculosis, or incompletely cured tuberculosis, as judged by the investigator and/or specialist (based on epidemiological history, symptoms, signs, laboratory tests, interferon-gamma release assay, imaging, etc.); unless there is documented evidence of adequate treatment or prophylactic anti-tuberculosis therapy started at least 2 weeks before the investigational product administration (and required to be used until the full course is completed), and the investigator and/or specialist judges that the subject can currently start JAK inhibitor treatment;
13. Chronic active infection or acute infection requiring systemic treatment with antibiotics, antiviral drugs, antiparasitic drugs, antiprotozoal drugs, or antifungal drugs within 4 weeks before screening; or superficial skin infection requiring treatment within 1 week before screening;
14. Known history of invasive infections (histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) (even if the infection has been resolved), or, in the investigator's judgment, abnormally frequent, recurrent, or prolonged infections suggesting possible immunodeficiency, or history of human immunodeficiency virus (HIV) infection;
15. Subjects with a history of thromboembolism (including deep vein thrombosis, pulmonary embolism, arterial thrombosis, etc.), or other high-risk populations prone to thromboembolism (the investigator comprehensively judges that such subjects are unsuitable for participation in this study based on clinical assessment);
16. Any of the following cardiovascular and cerebrovascular diseases/abnormalities:

    * Moderate to severe heart failure (New York Heart Association Class III or IV);
    * Previous large-area cerebral infarction/cerebral hemorrhage, myocardial infarction, coronary artery stent implantation;
    * Poorly controlled or refractory hypertension (after drug control, systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
    * Significant abnormalities on electrocardiogram (ECG), which, in the investigator's judgment, may pose an unacceptable risk to the subject participating in the clinical study, including but not limited to severe arrhythmia, QT interval corrected for heart rate using Fridericia's formula (QTcF) >480 ms;
    * Other cardiovascular and cerebrovascular-related medical histories/abnormalities that, in the investigator's judgment, make the subject unsuitable for participation in this study.
17. Subjects who have undergone or plan to undergo organ transplant surgery and require immunosuppressants (e.g., liver or kidney transplantation);
18. History of gastrointestinal perforation (except appendicitis or penetrating injury) or diverticulitis;
19. Conditions that may interfere with drug absorption, including but not limited to short bowel syndrome, gastrectomy, or specific types of bariatric surgery (e.g., gastric bypass surgery);
20. History of any malignancy, except successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix;
21. History of drug or alcohol abuse within 6 months before screening;
22. Other cardiovascular diseases, respiratory diseases, digestive diseases, endocrine diseases, autoimmune diseases, hematological diseases, urinary diseases, neuropsychiatric diseases, etc., that the investigator deems unsuitable for participation in this study;
23. Subjects who have undergone major surgery within 8 weeks before baseline or plan to undergo major surgery during the study period;
24. Blood loss ≥400 mL (including trauma, blood sampling, blood donation) within 12 weeks before baseline, or plan to donate blood during the study period or within 1 month after the study ends;
25. Inability to take oral tablets or allergy to the active ingredient or excipients of the investigational product;

    Have any of the following laboratory abnormalities:
26. Laboratory abnormalities during screening and at baseline:

    * Blood routine: white blood cells <2.5×10⁹/L, neutrophils <1.5×10⁹/L, lymphocyte count <0.8×10⁹/L; platelet count <100×10⁹/L, hemoglobin <100 g/L;
    * Renal function: estimated glomerular filtration rate (eGFR) <40 mL/min/1.73m², calculated using the Modification of Diet in Renal Disease (MDRD) formula;
    * Liver function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0× upper limit of normal (ULN) or total bilirubin (TBIL) >1.5×ULN;
    * Coagulation function: prothrombin time (PT) or activated partial thromboplastin time (APTT) >1.5×ULN;
27. Abnormalities during screening:

    * Hepatitis B surface antigen (HBsAg) positive; or hepatitis B core antibody (HBcAb) positive and hepatitis B virus deoxyribonucleic acid (HBV-DNA) positive;
    * Hepatitis C virus (HCV) antibody positive and hepatitis C virus ribonucleic acid (HCV-RNA) positive;
    * Human immunodeficiency virus (HIV) antibody positive;
    * Treponema pallidum antibody positive (except subjects with negative non-treponemal test results and judged by the investigator to have had past syphilis infection that has been cured); [Note] If a subject has abnormal laboratory test results during screening, the investigator may arrange one retest on a different day within the 35-day screening period (no drug intervention for the abnormal laboratory results is allowed before retesting), and the retest results will be used as the basis for determining the subject's eligibility.

    Other:
28. Any subject whom the investigator considers unsuitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-05-18 (Estimated); Study Completion 2027-07-19 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieved EASI-75 at week 16 of treatment. | At week 16 of treatment
The proportion of subjects who achieved vIGA-AD 0/1 with a reduction of ≥2 points from baseline at week 16 of treatment. | At week 16 of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- EnitiateBioPharma, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided